CLINICAL TRIAL: NCT00509743
Title: An Open-Label, Single-Dose Study to Assess the Effects of Age, Weight, and Body Composition on the Pharmacokinetic Profile, Safety, and Tolerability of Intravenous Diclofenac Sodium (DIC075V) in Adult Volunteers
Brief Title: Study to Assess Effects of Age, Weight, and Body Composition on the Pharmacokinetics of IV Diclofenac Sodium
Acronym: DFC-PK-008
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Javelin Pharmaceuticals (Industry)
Responsible Party: Gabrielle Poirier, Javelin Pharmaceuticals
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: DFC-PK-008
Record Dates: First submitted 2007-07-27; First posted 2007-07-31 (Estimated); Last update posted 2009-02-12 (Estimated); Status verified 2009-02

CONDITIONS: Healthy
Keywords: Adult volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Low dose Diclofenac
  Interventions: Drug: Intravenous diclofenac sodium (DIC075V)
- B (Experimental): High dose Diclofenac
  Interventions: Drug: Intravenous diclofenac sodium (DIC075V)

INTERVENTIONS:
Drug: Intravenous diclofenac sodium (DIC075V) — High dose Diclofenac
  Arms: B
Drug: Intravenous diclofenac sodium (DIC075V) — Low Dose Diclofenac
  Arms: A

SUMMARY:
The purpose of this study is to assess the effects of age, weight, and body composition on the pharmacokinetic profile, safety, and tolerability of intravenous diclofenac sodium (DIC075V) in adult volunteers.

DETAILED DESCRIPTION:
This study is an open label, single center, single-dose study to assess the effects of age, weight, and body composition on the pharmacokinetic profile, safety, and tolerability of intravenous diclofenac sodium (DIC075V) in adult volunteers. This study will be conducted in two cohorts. The first cohort of subjects will be selected based on body mass index (BMI) and weight criteria. The second cohort of subjects will be selected based on age.

ELIGIBILITY:
Inclusion Criteria:

* Adult volunteers over age 18

Exclusion Criteria:

* Known allergy or hypersensitivity to diclofenac, aspirin, or other NSAIDs or to any of the excipients of the study preparation
* History of previous and/or present cerebral hemorrhage, peptic ulceration, GI bleeding or any bleeding diathesis, positive for hepatitis B or hepatitis C or HIV antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
To assess the effects of age, weight, and body composition on the pharmacokinetic profile, safety, and tolerability of intravenous diclofenac sodium (DIC075V) in adult volunteers. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: D. Ronald Goldwater, MD, Principal Investigator — Parexel; William Gerson, D.O., Principal Investigator — Comprehensive Phase One
Locations (2):
- United States (2):
  - Comprehensive Phase One, Miramar, Florida
  - PAREXEL International, Baltimore, Maryland